CLINICAL TRIAL: NCT04137926
Title: Shanghai Mental Health Center
Brief Title: A Multicenter Study on the Diagnosis and Intervention of New Biomarkers on the Prodromal Stage of Alzheimer's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CRC2019ZD03
Record Dates: First submitted 2019-10-21; First posted 2019-10-24 (Actual); Last update posted 2021-09-23 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: AD, MCI due to AD and Normal Control
Who Masked: Investigator, Outcomes Assessor
Masking Description: In this study, the clinical researchers are responsible for the clinical diagnosis of the subjects and the diagnosis of senile plaques. The biological sample testing agency receives the blind coded samples. After the repeated testing, the data are handed over to the blind statistical experts for statistics. The statistical experts only obtain the grouping information and biological sample data, but do not know the specific diagnosis grouping, so as to ensure the accuracy of the statistical results. The results were analyzed by the researchers after the completion of the statistics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Alzheimer's disease (Experimental)
  Interventions: Diagnostic Test: MicRNAs battery
- MCI due to AD (Experimental)
  Interventions: Diagnostic Test: MicRNAs battery
- Normal Elderly (Experimental)
  Interventions: Diagnostic Test: MicRNAs battery

INTERVENTIONS:
Diagnostic Test: MicRNAs battery — for MCI due to AD diagnosis

SUMMARY:
The prevalence of Mild Cognitive Impairment (MCI) is about 15%-17%. 10%-15% of MCI progresses to Alzheimer's disease (AD) every year. The annual incidence of MCI in the normal elderly is about 1%. is the key and difficult points in AD research. Except expensive brain β amyloid plaque imaging, few breakthroughs of early diagnosis technology of MCI due to AD can be made to facilitate clinical application. The purpose of this program is to study the reliability and validity of plasma miRNAs for early diagnosis of MCI due to AD. The clinical diagnosis of AD and MCI due to AD are according to the National Institute of Aging and the Alzheimer's Disease Association (NIA-AA) diagnostic criteria in 2011. [18F]-AV-45 plaque imaging is used to be golden criteria for the diagnosis of AD and MCI due to AD. Next, a pilot intervention study on APP/PS1 transgenic mice will be promoted based on miRNAs gene regulation.

ELIGIBILITY:
Inclusion Criteria:

* 2011 NIA-AA criteria of MCI due to AD or AD

Exclusion Criteria:

* Non AD dementia

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
the diagnostic accuracy of biomarkers for MCI due to AD | 2 years
  MicRNAs battery for diagnostic of MCI due to AD
Neropsychological test battery | 2 years
  MicRNAs for intervene of MCI due to AD

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 years
  Number of participants with treatment-related adverse events as assessed by MicRNAs.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychogeriatrics，Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
After the study is finished.